CLINICAL TRIAL: NCT07274605
Title: Comparing the Therapeutic Efficacy of Extended Isthmusectomy Versus Total Thyroidectomy for Isthmus Tumors of the Thyroid: A Prospective, Multicenter, Open-Label, Randomized Controlled Trial.
Brief Title: Comparing the Therapeutic Efficacy of Extended Isthmusectomy Versus Total Thyroidectomy for Isthmus Tumors of the Thyroid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1245
Record Dates: First submitted 2025-11-24; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Thymectomy; Thyroid Cancer
Keywords: thyroid cancer; isthmus; surgery
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total thyroidectomy (Active Comparator): Patients randomised to this arm will undergo total thyroidectomy with bilateral central compartment (level VI) neck dissection
  Interventions: Procedure: Total thyroidectomy
- extended isthmusectomy (Experimental): Patients randomised to this arm will undergo extended isthmusectomy (ensure R0 resection) with bilateral central compartment (level VI) neck dissection
  Interventions: Procedure: Extended isthmusectomy

INTERVENTIONS:
Procedure: Total thyroidectomy — Total Thyroidectomy with bilateral central compartment (level VI) neck dissection - surgical removal of entire thyroid gland and perform bilateral Level VI neck dissection. This is the standard treatment recommended by the Chinese Guidelines for the Diagnosis and Management of Thyroid Nodules and Differentiated Thyroid Cancer (2nd Edition).
  The participating surgeons all routinely perform complete central neck dissections. They were selected for this study due to their standardized technique, which ensures a consistent surgical approach.
  Arms: Total thyroidectomy
Procedure: Extended isthmusectomy — Extended isthmusectomy with bilateral central compartment (level VI) neck dissection : Completely resect the isthmus and portions of the bilateral thyroid gland adjacent to the isthmus, ensuring an R0 resection margin for the tumor, while preserving at least more than half of the bilateral thyroid lobes.
  Arms: extended isthmusectomy

SUMMARY:
Prospective randomized open phase III non-inferiority trial in cT1bN0N1aM0 isthmus tumors of the thyroid comparing: extended Isthmusectomy (Isthmusectomy + Central Neck Dissection)(experimental group) versus total thyroidectomy + Central Neck Dissection (reference group).

DETAILED DESCRIPTION:
The thyroid isthmus is a narrow structure connecting the two lobes of the thyroid. Papillary carcinoma arising from this site accounts for only 1-9% of all thyroid cancers. However, due to its unique anatomical location, it is more prone to extranodal extension and bilateral lymph node metastasis, exhibiting more aggressive biological behavior. The optimal extent of surgery remains controversial: total thyroidectomy facilitates postoperative radioactive iodine therapy and monitoring but results in permanent dependence on thyroid hormone replacement and increases the risk of complications such as hypocalcemia, adversely affecting patients' quality of life. In contrast, conservative approaches like extended isthmusectomy can preserve partial thyroid function, reduce complications, and maintain a better quality of life, making them particularly suitable for low-risk patients with small tumors and no metastasis. Existing retrospective studies indicate no significant difference in recurrence rates between the two surgical approaches, though the evidence remains limited. Therefore, this study aims to conduct a prospective, multicenter, open-label, parallel-controlled, randomized trial to directly compare total thyroidectomy and extended isthmusectomy in terms of postoperative recurrence rates, quality of life, and complications, thereby providing high-quality evidence for surgical decision-making.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 years or older.

Diagnosis of low-risk differentiated thyroid cancer (papillary, follicular, or Hürthle cell carcinoma).

Unifocal tumor located in the thyroid isthmus, cT1b

No evidence of extrathyroidal extension, assessed by preoperative ultrasound.

Exclusion Criteria:

- Aggressive pathological subtypes (e.g., tall cell, clear cell, columnar cell, or diffuse sclerosing variants of papillary thyroid carcinoma, as well as poorly differentiated types).

cN1b.

M1

Combined with other suspicious thyroid nodules within the lobes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of 3-year recurrence | maximum of 3 years after the surgery
  defined as thyroid cancer recurrence, metastatic disease from thyroid cancer (whichever occurs first)

SECONDARY OUTCOMES:
Anatomical location of tumor recurrence | maximum of 3 years after the surgery
Risk of surgical site recurrence | maximum of 3 years after the surgery
  recurrence occured in the thyroid bed
Health Related Quality of Life | Baseline (post-randomisation/pre-surgery), 4 weeks and 3, 6,12 months after the surgery
  Measured using FoP-Q-SF: Scales range from 12-60 with higher scores indicating greater fear of disease progression Measured using THYCA-Qol questionnaires: including 7 symptom dimensions and 6 single items. All items are rated on a 4-point scale (none, a little, quite a bit, very much), scored from 1 to 4. Higher scores on individual items indicate lower quality of life.
Number of participants with Hormone Replacement Therapy | 2-4 weeks and 3, 6, 12, 24, 36 months after the surgery
  patients who require thyroxin intake
Rate of surgical complications | perioperatively, 2-4 weeks, 6 months after the surgery
  including transient/permanent hypoparathyroidism, transient/permanent recurrent laryngeal nerve injury, postoperative infection, and postoperative lymphatic fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyu Li, MD, Principal Investigator — Thyroid surgery Department, 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided